CLINICAL TRIAL: NCT05995470
Title: Effect of an Internet-based Dialectical Behaviour Therapy-informed Skills Training for Reducing Alcohol Consumption and Improving Psychological Distress of Adult Drinkers: A Pilot Randomised Controlled Trial
Brief Title: Effect of an Internet-based Dialectical Behaviour Therapy-informed Skills Training for Adult Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ho Long Kwan, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07210047
Record Dates: First submitted 2023-08-02; First posted 2023-08-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Drinking
Keywords: Dialectical behaviour therapy; Skills training; Internet-based intervention; Psychological distress; Alcohol drinking; Adult drinkers
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBT-ST group (Experimental): Participants in the intervention group will receive the DBT-ST by means of a free video-communication app. Over the next 13 weeks from the baseline, the intervention group will receive a weekly 120-minute internet-based DBT-ST focusing on the four modules of DBT-ST.
  Interventions: Behavioral: Internet-based dialectical behaviour therapy-informed skills training
- TAU group (Other): Participants in the wait list control group will receive a monthly health education for three months that provides general health information and sharing sessions, which is one of the routine care for drinkers during the first 3-4 months after they seek help for drinking problem (waiting period for further intervention).
  Interventions: Behavioral: Monthly health education

INTERVENTIONS:
Behavioral: Internet-based dialectical behaviour therapy-informed skills training — Adaptive applications of DBT-ST for drinkers with psychological distress
  Arms: DBT-ST group
Behavioral: Monthly health education — General health information and sharing sessions
  Arms: TAU group

SUMMARY:
1. To determine the feasibility, acceptability, and preliminary effects of an internet-based DBT-ST for reducing alcohol consumption and improving psychological distress/emotional regulation in adult drinkers
2. To explore the participants' experiences and perceptions of the proposed intervention

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese aged ≥18
* Score ≥8 on the Alcohol Use Disorders Identification Test
* Indicate psychological distress as measured by the Depression, Anxiety, and Stress Scale-21
* Have an intention to stop drinking
* Have an electronic device and are willing to receive interventions via the internet

Exclusion Criteria:

* Experiencing psychotic disorders/cognitive impairment/communication problems
* Participating in other alcohol abstinence/related psychosocial interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-01-21 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption | Baseline, Post-intervention (upon completion of the 13-week DBT-ST), 3-month post-intervention
  The Chinese version of the Alcohol Use Disorders Identification Test-Concise (AUDIT-C)
Level of psychological distress | Baseline, Post-intervention (upon completion of the 13-week DBT-ST), 3-month post-intervention
  Symptoms of depression, anxiety and stress

SECONDARY OUTCOMES:
Self-reported alcohol abstinence | Baseline, Post-intervention (upon completion of the 13-week DBT-ST), 3-month post-intervention
  Self-reporting of quitting
Emotion dysregulation | Baseline, Post-intervention (upon completion of the 13-week DBT-ST), 3-month post-intervention
  Levels of emotion dysregulation
Distress tolerance | Baseline, Post-intervention (upon completion of the 13-week DBT-ST), 3-month post-intervention
  Perceived ability to tolerate emotional distress
Coping response | Baseline, Post-intervention (upon completion of the 13-week DBT-ST), 3-month post-intervention
  Self-report measure of coping strategies

OTHER OUTCOMES:
Acceptability | Post-intervention (upon completion of the 13-week DBT-ST)
  Client Satisfaction
Feasibility of the intervention | Post-intervention (upon completion of the 13-week DBT-ST)
  1) Recruitment rate; (2) Intervention engagement in terms of time spent on each session and participation rates; and (3) Attrition rates
Semi-structured interview | Post-intervention (upon completion of the 13-week DBT-ST)
  Individual semi-structured interviews will be conducted at post-intervention to explore participants' experiences/perceptions of the internet-based DBT-ST, as well as their comments on the appropriateness/comprehensiveness of the content/frequency of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Long Kwan Ho, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Hospital Authority, Hong Kong, Hong Kong